CLINICAL TRIAL: NCT01772940
Title: Nevirapine vs Ritonavir-boosted Lopinavir in ART HIV-infected Adults in a Resource-limited Setting; a Randomized, Multicenter, Parallel Group Study
Brief Title: Nevirapine vs Ritonavir-boosted Lopinavir in ART Naive HIV-infected Adults in a Resource Limited Setting
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Saint Pierre (Other)
Collaborators: University of Liege (Other); Ministry of Public Health, Democratic Republic of the Congo (Other Government); Pierre and Marie Curie University (Other); University Paris 7 - Denis Diderot (Other); Gilead Sciences (Industry); Abbott (Industry)
Responsible Party: Principal Investigator, Clumeck Nathan, Chief infectious diseases , Professor of Medicine, Centre Hospitalier Universitaire Saint Pierre
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: Lubumbashi trial
Record Dates: First submitted 2013-01-14; First posted 2013-01-21 (Estimated); Last update posted 2013-08-26 (Estimated); Status verified 2013-08

CONDITIONS: HIV-1 Infection
Keywords: First-line therapy; Protease inhibitor; Non-Nucleoside Reverse transcriptase Inhibitor; Resource-limited setting
MeSH Terms: interventions — Nevirapine; lopinavir-ritonavir drug combination; Tenofovir; Emtricitabine; Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination; lamivudine, zidovudine drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- nevirapine and tenofovir/emtricitabine (Active Comparator): nevirapine 200 mg twice daily combined with tenofovir 300 mg/emtricitabine 200 mg (fixed-dose combination) once daily, per os for 96 weeks
  Interventions: Drug: nevirapine; Drug: Tenofovir/emtricitabine
- lopinavir/r and tenofovir/emtricitabine (Experimental): ritonavir-boosted lopinavir 800/200 mg once daily or 400/100 mg twice daily combined with tenofovir 300 mg/emtricitabine 200 mg (fixed-dose combination) once daily, per os for 96 weeks
  Interventions: Drug: ritonavir-boosted Lopinavir; Drug: Tenofovir/emtricitabine
- Nevirapine and zidovudine/lamivudine (Active Comparator): nevirapine 200 mg/zidovudine 300 mg/lamivudine 150 mg (fixed-dose combination) twice daily, per os for 96 weeks
  Interventions: Drug: nevirapine; Drug: Zidovudine/lamivudine
- Lopinavir/r and zidovudine/lamivudine (Experimental): ritonavir-boosted lopinavir 800/200 mg once daily or 400/100 mg once daily combined with zidovudine 300 mg/lamivudine 150 mg once daily, per os for 96 weeks
  Interventions: Drug: ritonavir-boosted Lopinavir; Drug: Zidovudine/lamivudine

INTERVENTIONS:
Drug: nevirapine — Nevirapine 200 mg twice daily or 400 mg once daily per os during 96 weeks
  Other Names: Viramune
  Arms: Nevirapine and zidovudine/lamivudine; nevirapine and tenofovir/emtricitabine
Drug: ritonavir-boosted Lopinavir — ritonavir-boosted lopinavir 800/200 mg once daily or 400/100 mg twice daily per os during 96 weeks
  Other Names: Aluvia
  Arms: Lopinavir/r and zidovudine/lamivudine; lopinavir/r and tenofovir/emtricitabine
Drug: Tenofovir/emtricitabine — tenofovir 300 mg/emtricitabine 200 mg fixed-dose combination once daily, per os for 96 weeks
  Other Names: Truvada
  Arms: lopinavir/r and tenofovir/emtricitabine; nevirapine and tenofovir/emtricitabine
Drug: Zidovudine/lamivudine — zidovudine 300 mg/lamivudine 150 mg twice daily fixed-dose generic combination, per os for 96 weeks
  Other Names: Zidolam,combivir
  Arms: Lopinavir/r and zidovudine/lamivudine; Nevirapine and zidovudine/lamivudine

SUMMARY:
In resource-limited setting, concerns remain regarding the emergence of virologic failure and high-level drug resistance mutations (DRM) during WHO recommended first-line antiretroviral therapy (ART) with non-nucleoside reverse transcriptase inhibitors (NNRTI) based regimens for Human immunodeficiency virus 1 (HIV1) infected patients. The study hypothesis is that a boosted-protease inhibitor regimen has a better outcome than a NNRTI-based regimen with a low genetic barrier to resistance.

The study is a randomized, multicenter, factorial trial (conducted in Congo), in treatment- naïve adults receiving for 96 weeks ritonavir- boosted lopinavir(LPV/r) or nevirapine (NVP) each in combination with tenofovir (TDF) /emtricitabine (FTC) or zidovudine (ZDV)/lamivudine (3TC). The primary end point is the incidence of therapeutic (clinical and/or virologic)failure by study week 24.

ELIGIBILITY:
Inclusion Criteria:

* Antiretroviral-therapy naïve HIV-1 infected Adults
* WHO clinical stage 3 and CD4 <350/mm3 or
* WHO clinical stage 4 or
* CD4 cell count < 200/mm3
* Negative pregnancy test

Exclusion Criteria:

* Hemoglobin < 8.5 g/dL (female) or 9.0 g/dL (male)
* Estimated Glomerular Filtration Rate < 50 ml/ minute (Cockcroft-Gault equation)
* Hepatic transaminases (AST and ALT)> 3 x upper limit of normal
* Active tuberculosis
* Pregnancy
* Females who are breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 425 (Actual)
Dates: Start 2008-12; Primary Completion 2011-10 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Incidence of therapeutic failure | At week 48 with follow-up until week 96
  The primary end point is the proportion of patients with therapeutic failure defined as:
  * the occurence or relapse by week 24 of a World Health Organization (WHO) stage 4 or 3 event, or
  * death by week 24, or
  * discontinuation of study drugs due to toxicity at any time, or
  * virological failure defined as HIV-1 RNA > 1000 copies/ml by week 24

SECONDARY OUTCOMES:
HIV-1 RNA viral load less than 50 copies/ml | Through week 96
  The percentage of patients with HIV-1 RNA < 50 copies/ml
Immunologic response | Through week 96
  Cluster of differentiation 4 (CD4) cell count change from baseline
HIV-1 resistance mutations | At baseline and at the time of virologic failure
Safety and tolerability | Through week 96
  Incidence of adverse events and laboratory abnormalities
Changes in laboratory parameters | Through week 96

CONTACTS AND LOCATIONS:
Overall Officials: Nathan Clumeck, MD, PhD, Principal Investigator — Centre Hospitalier Universitaire Saint Pierre
Locations (1):
- Cliniques Universitaires de Lubumbashi, Lubumbashi, Katanga, Republic of the Congo

REFERENCES:
- [Derived] Clumeck N, Mwamba C, Kabeya K, Matanda S, Vaira D, Necsoi C, Kadiebwe D, Delforge M, Kasamba E, Milolo C, Ilunga J, Kapend L. First-line antiretroviral therapy with nevirapine versus lopinavir-ritonavir based regimens in a resource-limited setting. AIDS. 2014 May 15;28(8):1143-53. doi: 10.1097/QAD.0000000000000214. PMID 25028911